CLINICAL TRIAL: NCT04198675
Title: Effects of Preventive Physiotherapy Practices on Forward Head Posture and Upper Extremity Work-Related Functions in Office Workers
Brief Title: Effects of Preventive Physiotherapy Practices on Posture and Work-Related Functions in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Nilufer Keskin Dilbay, PT, MSc, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09.2018.282
Record Dates: First submitted 2019-09-01; First posted 2019-12-13 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Work-related Musculoskeletal Disorders; Office Workers
Keywords: Surface Electromyography; Biofeedback; Forward Head Posture; Posture; Trapezius Muscle; Task- specific Performance; Exercise; Office Worker
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Group 1: Supervised EMG Biofeedback Exercise Training Group; Posture training will be provided before intervention and ergonomic arrangements will be made in the workplace. Three sessions per week and six weeks of EMG biofeedback training will be carried out with electromyography-controlled video game combined with Proprioceptive Neuromuscular Facilitation (PNF) exercises.
  Group 2: Home-Based Exercise Training Group; Posture training will be provided before interventions and ergonomic arrangements will be made in the workplace. Posture correction exercises, contains strengthening, stretching, mobility and relaxation exercises, will be given as a home exercises program for 6 weeks.
  Group 3: Posture Training/Ergonomic Regulations Group Posture training will be provided before interventions and ergonomic arrangements will be made in the workplace.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised EMG Biofeedback Exercise Training Group (Active Comparator): Frequency: 3/week Duration:6 weeks Dosage: Tolerable intensity-dependent increase in exercises program.
  Interventions: Behavioral: Supervised EMG Biofeedback Exercise Training Group
- Home-Based Exercise Training Group (Active Comparator): Frequency: 3/week Duration:6 weeks Dosage: Tolerable intensity-dependent increase in exercises program.
  Interventions: Behavioral: Home-Based Exercise Training Group
- Posture Training/Ergonomic Regulations Group (Sham Comparator): 1 session, no further intervention until second evaluation for 6 weeks.
  Interventions: Behavioral: Posture Training/Ergonomic Regulations Group

INTERVENTIONS:
Behavioral: Supervised EMG Biofeedback Exercise Training Group — Posture training and ergonomic arrangements in the workplace. EMG biofeedback training will be carried out with electromyography-controlled video game combined with PNF exercises. Each game sessions comprising the work-rest cycle covers performing the upper trapezius muscle contraction simultaneously the upper extremity PNF patterns.
  Arms: Supervised EMG Biofeedback Exercise Training Group
Behavioral: Home-Based Exercise Training Group — Posture training and ergonomic arrangements in the workplace. Posture correction exercises, contains strengthening, stretching, mobility and relaxation exercises, will be given as a home exercises program. Exercise diary and weekly calls will be use to maintain the exercise adherence
  Arms: Home-Based Exercise Training Group
Behavioral: Posture Training/Ergonomic Regulations Group — Posture training and ergonomic arrangements in the workplace.
  Arms: Posture Training/Ergonomic Regulations Group

SUMMARY:
In this study; aimed to determine an individual-centered, effective physiotherapy method to reduce the negative impacts of the forward head posture on work-related functions and to increase body awareness and functionality among office workers. In addition, aimed to reduce the loss of work with measures to improve the quality and efficiency of work.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of preventive physiotherapy practices on work related musculoskeletal disorders in office workers.

With this purpose, in this study; aimed to achieve improvement on forward head posture, upper extremity functions and cervical pain reduction through three interventions (supervised EMG biofeedback exercise training, home-based exercise program and posture training/ergonomic regulations). Work related changes in muscle activation of Upper Trapezius and posture will be evaluated while working on a computer task in actual work environment. Differences in posture and muscle activation between computer task and resting position, will be determined before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age below 40, Full-time and regular employees in the last 1 year,
* Office workers using computers at desk for at least 3 hours per day
* According to RULA, working in a posture that above acceptable level,
* No trauma history
* Non-specific neck pain but no chronic conditions of cervical spine and upper extremity

Exclusion Criteria:

* During the study; need of receiving a treatment/ interventions for the upper body due to trauma or any other conditions is concluded with withdraw from the study

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction (MVIC) | 10 minutes
  It is assessed by Surface Electromyography (sEMG) for upper trapezius muscle. 3 maximum contractions are performed for 6 seconds at the manual muscle testing position. The maximum value among 3 repeats is recorded as Maximal Voluntary Isometric Contraction (MVIC) (mV).
Muscle Activation of Upper Trapezius | 30 minutes
  It is the measurement of the Electromyographic activity of trapezius muscles during functional tasks and rest. According to The Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles Project (SENIAM) recommendations for sensors and sensor placement procedures, sEMG will be applied for the upper trapezius muscles while resting and also performing the computer task in workplace. The mean values (mV) obtained are normalized according to MVIC. Normalized data (%MVIC) are used in the statistical analysis.
Cervical Range of Motion (CROM) / Forward Head Posture | 10 minutes
  The CROM Deluxe is an assessment instrument that lets to measure sagittal, frontal and horizontal plane movements (flexion / extension, lateral flexion, rotation and forward head posture), while resting and also performing a task or work posture.

SECONDARY OUTCOMES:
Constant-Murley Score (CMS) | 10 minutes
  The Constant-Murley Score (CMS) is a widely used scale to measure pain, mobility and the ability to carry out the normal daily activities in various shoulder conditions/ pathologies.
Rapid Upper Limb Assessment (RULA) | 10 minutes
  The RULA Assessment Tool is used to evaluate the ergonomic risk factors associated with neck, trunk and upper extremity Musculoskeletal Disorders (MSD). The RULA considers biomechanical and postural load requirements of job demands. Scores between 1-7 are classified from "acceptable posture" (no action required) to "very high risk" (implement change now).
The Disabilities of the Arm, Shoulder and Hand Score (DASH) | 10 minutes
  The DASH is a self reported questionnaire; assesses the parameters of daily life, pain, weakness, social functions, work, sleep and self-confidence associated with the upper extremity of the individual.
The Disabilities of the Arm, Shoulder and Hand Score Work Module (DASH-W) | 2 minutes
  Work Module (DASH-W) is the second part of the DASH questionnaire, which consists of 4 questions, determines one's disability in working life.
Neck Disability Index (NDI) | 10 minutes
  The NDI is a self-reported scale consists of pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping and leisure time activities sections. The total score varies between 0-50 and the increase in total score indicates the increase in the severity of the neck disability.
Neck Pain and Disability Scale (NPAD) | 10 minutes
  The NPAD is a self-reported index which measure the intensity of neck pain during different conditions and activities and related effects of pain on occupational, recreational, social, daily living activities and its relationship with emotional factors. Pain-related data are obtained by marking on visual analogue scales of 20 items.

CONTACTS AND LOCATIONS:
Overall Officials: Nilufer Keskin Dilbay, PT, MSc, Principal Investigator — Marmara University; Zafer Erden, PT PhD Prof., Study Director — Hacettepe University
Locations (1):
- Marmara University Faculty of Health Sciences, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No